CLINICAL TRIAL: NCT01011777
Title: Phase I Study of Endoscopically Injected Muscle Derived Cells in Participants With Exstrophy-epispadias Complex Related Urinary Incontinence
Brief Title: Muscle Derived Cell Therapy for Bladder Exstrophy Epispadias Induced Incontinence
Acronym: MDC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to participants withdrawal prior to anticipated end of study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061692
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Bladder Exstrophy; Urinary Incontinence
Keywords: bladder exstrophy epispadias complex; urinary incontinence; muscle derive cell therapy; stem cells
MeSH Terms: conditions — Bladder Exstrophy; Urinary Incontinence; Bladder Exstrophy and Epispadias Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Muscle Derived Cells (Experimental): Surgeon will endoscopically inject previously harvested autologous muscle derived cells (MDC) into the same bladder exstrophy patient's urinary sphincter to improve outflow resistance and rhabdosphincter contractility. We will assess tolerability and induction of continence.
  Interventions: Drug: MDC

INTERVENTIONS:
Drug: MDC — After the biopsy the MDC expansion process takes approximately 21 days after which cells are harvested and cryopreserved for future injection. The MDC product is stored in single use vials, with each vial containing approximately 2.6 x 10^7 total cells. The volume of each vial will be 1.3ml. This study uses a single dose of approximately 2.0 x 10^7 cells administered endoscopically into the external urethral sphincter in 12 injections of 0.1ml each. Six months post-initial MDC injection, group 1 participants with persistent bladder capacity less than 100cc and group 2 participants with persistent urinary incontinence as defined in eligibility criteria may undergo repeat injections of MDC at 6 month intervals for up to a total of 4 injections.
  Other Names: Autologous Muscle Derived Cells

SUMMARY:
The aim of this study is to study safety, tolerability and efficacy of muscle derived cell (MDC) therapy in children with bladder exstrophy epispadias induced urinary incontinence.

DETAILED DESCRIPTION:
Bladder exstrophy patients who have undergone primary bladder closure, but have a bladder capacity too low for bladder neck reconstruction (Group 1), have limited additional surgical options that permits urethral voiding and urine storage within a native bladder. Previous studies have demonstrated a positive correlation between bladder capacity and success of bladder neck reconstruction. Likewise, patients who have undergone bladder neck reconstruction but continue to have urinary incontinence (Group 2) are also faced with limited options. Often, both groups are considered for augmentation cystoplasty with closure of the bladder neck requiring intermittent catheter voiding through a surgically constructed continent catheterizable channel. Such major reconstruction has significant associated short and long-term morbidities. Endoscopic injection of MDCs for the treatment of urinary sphincter insufficiency is a potential alternative therapy for these patients. By increasing the outflow resistance and rhabdosphincter contractility, MDC injection may permit more efficient bladder cycling and bladder expansion in Group 1 patients allowing them to proceed on to bladder neck reconstruction. This same increase in resistance and sphincter contractility may allow Group 2 patients to attain urinary continence and avoid any further reconstructive surgical procedures.

Eligible and consented patients would undergo rectus muscle biopsy and immediately transferred to the Cell Therapy Lab for tissue processing and MDC expansion.The MDC expansion process takes approximately 21 days after which cells are harvest and cryopreserved for future injection.Each vial will be filled with cells at a concentration of approximately 2.0 x 107 cells/ml. At the time of planned MDC injection, enrolled patients will return for cystoscopy under anesthesia. At that time, aliquots of MDCs will be removed from the freezer and be allowed to thaw passively in the 30 minutes preceding the time of planned injection. MDC product will be endoscopically injected using an FDA approved DEFLUX™ needle at the level of the external urethral rhabdosphincter and bladder neck. Patients would be assessed for toxicity and adverse events postoperatively at day 1 and 40 followed by semiannual visits for 36 months. variables measured are:

group 1: Bladder capacity, detrusor leak point pressure, bladder filling pressure, post-void residual urine volume, urodynamics, periurethral electromyographic activity, renal - Bladder Ultrasound, cystoscopy.

Group 2: Detrusor leak point pressure, bladder filling pressure, maximum cystometric capacity, post-void residual urine volume, periurethral electromyographic activity, 24 hour pad / diaper weight assessment, voiding diary including incontinence grade and maximum daytime dry interval, renal - Bladder Ultrasound, cystoscopy

ELIGIBILITY:
Inclusion Criteria:

1. Group 1 - Males and females at least 2 years of age with:

   * Classic bladder exstrophy with successful primary, secondary, or delayed primary closure and subsequent epispadias repair.
   * Cystography done with 90 days preceding participant identification and at least 12 months after successful bladder closure demonstrating a bladder capacity less than 100cc.
2. Group 2 - Males and females greater than 5 years of age with:

   * Classic bladder exstrophy with successful primary, secondary, or delayed primary closure and subsequent epispadias repair.
   * Previous bladder neck reconstruction.
   * At the time of participant identification, urinary incontinence defined as leakage of urine at night or leakage of urine at an interval of less than 3 hours in the daytime persisting at least 2 years after bladder neck reconstruction.
3. Screening labs obtained less than 30 days prior to MDC injection meeting the following criteria:

   * Urinalysis and urine culture demonstrating either no bacterial growth or growth of an organism that can be treated with an appropriate oral antibiotic for 7 days preoperatively. Participants with a positive urine culture should have the urinalysis and urine culture repeated after completion of antibiotics and prior to MDC injection. A negative urine culture must be demonstrated prior to MDC injection.
   * Serum creatinine in normal range for age (Infant: 0.2-0.4 mg/dl; Child 0.3-0.7 mg/dl; Adolescent 0.5-1.0 mg/dl).
   * Negative Study Donor Virology Panel (Hep B surface antigen, HIV 1 / 2 antibody, Hep B core antibody, Rapid Plasma Reagin (RPR), Human T-cell Lymphotrophic Virus (HTLV) I / II antibody, Hep C antibody). This panel is only done during the screening process and is not repeated during study follow-up.
4. Parent or legal guardian who is, in the opinion of the investigator, reliable and willing to make themselves and patient available for the duration of the study and are willing to follow study procedures and unit policies.
5. Parent or legal guardian able to complete and sign the informed consent document.
6. Negative pregnancy test for sexual active female teenagers. If able to conceive and sexually active, participants must agree to use barrier contraceptives from the time of study enrollment until 6 months after the last MDC injection. Male participants who are able to conceive and are sexually active must agree to use protection as well from the time of study enrollment until 6 months after the last MDC injection.

Exclusion Criteria:

1. Urodynamic study demonstrating severe uninhibited bladder contractions.
2. Severe urethral or bladder neck stricture demonstrated during screening cystoscopy or cystogram
3. Cystography at the time of screening demonstrating Grade IV vesicoureteral reflux (high-grade reflux with dilation of the renal pelvis and blunting or the fornices) or Grade V vesicoureteral reflux (Grade IV findings plus loss of the papillary impression and ureteral tortuosity).
4. Any degree of renal scarring at the time of screening as demonstrated by DMSA or MAG3 renal scintigraphy in the presence of any grade of vesicoureteral reflux (VUR)
5. Renal ultrasound demonstrating Society of Fetal Urology Grade III hydronephrosis (widely split renal pelvis, renal calices uniformly dilated, no parenchymal thinning) or Grade IV hydronephrosis (Grade III dilation plus parenchymal thinning). See Appendix D.
6. Previous injection of bulking agents at the level of the bladder neck (bovine collagen or DEFLUX™)
7. Positive urine culture resistant to preoperative oral antibiotic therapy
8. Need for chronic or pulse steroids or history of other congenital or acquired condition that results in immunocompromise
9. Previous adverse reaction to anesthesia

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
The ability to inject the MDC product in a safe and tolerable manner in a clinical setting using a descriptive approach. | Post op day 1, day 40, monthly afterwards for 36 months

SECONDARY OUTCOMES:
changes in urinary incontinence levels and bladder growth in enrolled participants after undergoing autologous MDC injection using cystograms, urodynamic studies, 24-hour pad weight test, continence score, and maximum day & nighttime dry interval. | Monthly voiding diary. All other parameters measure at baseline and every 6 months for 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: John P Gearhart, MD, Principal Investigator — Brady Urological Institute, Department of Pediatric Urology
Locations (1):
- Brady Urological Institute. Johns Hopkins University, Baltimore, Maryland, United States